CLINICAL TRIAL: NCT05334758
Title: Clinical Performance Evaluation of the Bio-Self™ COVID-19 Antigen Home Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTeke USA, LLC (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BTK-01-1002
Record Dates: First submitted 2022-04-15; First posted 2022-04-19 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: Covid, Covid 19, Virus
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective study to evaluate the sensitivity and specificity of the Bio-Self COVID-19 Antigen Home Test when a lay person conducts the test on themselves or another study participant. Potential subjects will be those presenting for COVID-19 testing. The study will evaluate the performance of the Bio-Self COVID-19 Antigen Home Test by comparing it to a high sensitivity EUA SARS-CoV-2 RT-PCR assay to calculate both the positive percent agreement [(PPA) sensitivity] and negative percent agreement [(NPA) specificity].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- At least 30 children between 2 - 13 years of age (Experimental): Subjects less than 14 years of age, where the Parent or legal guardian collects a sample from their child (e.g., ages 2-13) and performs the Bio-Self COVID-19 antigen home test. The standard of care test and the RT-PCR test samples will be collected by the study team.
  Interventions: Device: Bio-Self COVID-19 Antigen Home Test; Device: Standard of Care COVID-19 Test; Diagnostic Test: RT-PCR Test
- Subjects 14 - 90 years of age (Experimental): The subject will self collect and test using the Bio-Self COVID-19 antigen home test. The standard of care test and the RT-PCR test samples will be collected by the study team.
  Interventions: Device: Bio-Self COVID-19 Antigen Home Test; Device: Standard of Care COVID-19 Test; Diagnostic Test: RT-PCR Test

INTERVENTIONS:
Device: Bio-Self COVID-19 Antigen Home Test — At home COVID-19 antigen test kit
Device: Standard of Care COVID-19 Test — Standard of care
Diagnostic Test: RT-PCR Test — High Sensitivity RT-PCR COVID-19 Test

SUMMARY:
The purpose of this study is to evaluate the performance of the Bio-Self COVID-19 Antigen Home Test. The study will evaluate the accuracy (sensitivity and specificity) in a simulated home use environment when compared to a high-sensitivity Emergency Use Authorization (EUA) SARS-CoV-2 RT-PCR assay.

DETAILED DESCRIPTION:
The Bio-Self COVID-19 Antigen Home Test is immunochromatographic and uses double-antibody sandwich method to detect SARS-CoV-2 antigen from individuals with or without symptoms or other epidemiological reasons to suspect a COVID-19 infection. The test is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older or adult collected anterior nares swab samples from individuals ages 2 to 13.

The primary objective of this study is to determine the accuracy of the Bio-Self COVID-19 Antigen Home Test when compared to a high-sensitivity Emergency Use Authorization (EUA) SARS-CoV-2 RT-PCR assay.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent and assent, if applicable, is signed and dated prior to any study-related activities.
2. Male and female Subjects 2 years of age and older.
3. Subject is willing to provide a self-collected nasal swab sample. (If under the age of 14, the sample will be collected by an adult.)
4. Subject is willing to have a nasal swab collected by a healthcare professional.
5. Subject agrees to complete all aspects of the study.

Exclusion Criteria:

1. Subject has a visual impairment that cannot be restored with glasses or contact lenses.
2. Subject has prior medical or laboratory training.
3. Subject had a positive COVID-19 test in past three (3) months.
4. Subject uses home diagnostics, e.g., HIV Tests, glucose meters, etc.

Ages: 2 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Geller, MD, Principal Investigator — Centennial Medical Group; Enrique Villa, MD, Principal Investigator — L&A Morales Healthcare; Narendra Kini, MD, Principal Investigator — CDR Health
Locations (3):
- United States (3):
  - L&A Morales Healthcare, Inc., Miami, Florida
  - CDR Health, Tallahassee, Florida
  - Centennial Medical, Elkridge, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of First Enrollment: 12 May 2022 Date of Last Completed: 25 July 2022
  The first 50 subjects presenting to the sites for COVID-19 testing were consecutively enrolled (i.e., all comers) including those who were either asymptomatic or symptomatic for COVID-19. Following this enrollment, only subjects who were symptomatic for COVID-19 were enrolled until 30 RT-PCR confirmed positive samples were collected. Then enrollment resumed for all comers.
Period: Overall Study
Arm/Group | At Least 30 Children Between 2 - 13 Years of Age | Subjects 14 - 90 Years of Age
Started | 30 | 252
Completed | 30 | 252
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Performance analysis was based on 253 subjects rather than the 282 enrolled due to loss of samples. See Arm/Group Description for more details.
Groups:
- Performance Data Set: In the initial PEUA, the Agency confirmed that the EUA authorized high-sensitivity PerkinElmer New Coronavirus Nucleic Acid Detection Kit was an acceptable RT-PCR comparator for this study. In a follow-up email to the Agency on 18 July 2022, BioTeke asked if the chosen PerkinElmer RT-PCR kit could be utilized with a separately authorized extraction method (i.e., ThermoFisher KingFisher), which had been internally validated by the CLIA laboratory but was not included in the PerkinElmer's Instructions for Use. Of note, the initial subject samples had been tested using this extraction kit. The FDA responded that this would not be an acceptable approach, as the comparator method had to use the authorized extraction method outlined in the manufacturer's authorized instructions. In response to the Agency's decision, the central CLIA testing laboratory, DevLab Bio, internally validated the extraction method using the Chemagic 360 as specified in the PerkinElmer instructions. The intent was to re-test those samples previously tested using the ThermoFisher extraction method and test all future samples using only this authorized process.
  When preparing to re-test the initial subject samples, it was found that a number of samples had been discarded in error. These samples were not included in the performance analysis.
  Performance analysis was based on 253 subjects rather than the 282 enrolled.
Arm/Group | Performance Data Set
Number analyzed (Participants) | 253
Age, Customized [Count of Participants; unit: Participants]
  Age: < 14 years | 27
  Age: 14 - 24 years | 24
  Age: 25 - 64 years | 108
  Age: ≥ 65 years | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 132
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 222
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 253
Symptomatic [Count of Participants; unit: Participants] | 155

OUTCOME MEASURES:

1. Primary Outcome: Positive Percent Agreement - Sensitivity
Description: The sensitivity is computed as the proportion of positive samples as called by the EUA SARS-CoV-2 RT-PCR assay, which are also positive as called by the Bio-Self COVID-19 Antigen Home Test.
Time Frame: 48 hours
Population: Symptomatic Subjects
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- Performance Data Set: In the initial PEUA, the Agency confirmed that the EUA authorized high-sensitivity PerkinElmer New Coronavirus Nucleic Acid Detection Kit was an acceptable RT-PCR comparator for this study. In a follow-up email to the Agency on 18 July 2022, BioTeke asked if the chosen PerkinElmer RT-PCR kit could be utilized with a separately authorized extraction method (i.e., ThermoFisher KingFisher), which had been internally validated by the CLIA laboratory but was not included in the PerkinElmer's Instructions for Use. Of note, the initial subject samples had been tested using this extraction kit. The FDA responded that this would not be an acceptable approach, as the comparator method had to use the authorized extraction method outlined in the manufacturer's authorized instructions. In response to the Agency's decision, the central CLIA testing laboratory, DevLab Bio, internally validated the extraction method using the Chemagic 360 as specified in the PerkinElmer instructions. The intent was to re-test those samples previously tested using the ThermoFisher extraction method and test all future samples using only this authorized process.
  When preparing to re-test the initial subject samples, it was found that a number of samples had been discarded in error. These samples were not included in the performance analysis.
Arm/Group | Performance Data Set
Number analyzed (Participants) | 155
percent probability | 96.2 [87.2 to 99]

2. Primary Outcome: Negative Percent Agreement - Specificity
Description: The specificity is computed as the proportion of negative samples as called by the EUA SARS-CoV-2 RT-PCR assay, which are also negative as called by the Bio-Self COVID-19 Antigen Home Test.
Time Frame: 48 hours
Population: Specificity for symptomatic subjects
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Performance Data Set
Number analyzed (Participants) | 155
percent probability | 100 [96.4 to 100]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: This study was deemed to have a less than significant risk by IRB assessment, and no sites reported any adverse events during or after the study enrollment period.
Arm/Group | At Least 30 Children Between 2 - 13 Years of Age | Subjects 14 - 90 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/252
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/252
Other Adverse Events (participants affected / at risk) | 0/30 | 0/252

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT05334758/Prot_SAP_000.pdf